CLINICAL TRIAL: NCT05371184
Title: Safety and Efficacy of Glutamine in Preventing Vaso-occlusive Crisis Among Sickle Cell Disease Patients: Randomized Controlled Study
Brief Title: Glutamine Role in Preventing Vaso-occlusive Crisis Among SCD Patients
Acronym: Glu_SCD_Egy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma Soliman Elsayed Ebeid, MD, professor of pediatric hematology ,oncology and bone marrow transpalnt, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMASU MD 199/ 2021
Record Dates: First submitted 2022-05-04; First posted 2022-05-12 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Sickle Cell Disease
Keywords: glutamine, vasooclussive crisis, sickle cell disease, Egypt
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Glutamine; Powders; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cases (Experimental): • 30 patients will receive glutamine in a dose of 0.3 gm /kg/dose twice daily orally (up to a maximum of 15 g/dose) for 24 weeks as an add on to the SOC
  Interventions: Drug: L-Glutamine, Oral Powder for Reconstitution
- control (Active Comparator): 30 patients will be assigned as a control group to receive standard of care therapy without glutamine intake.
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: L-Glutamine, Oral Powder for Reconstitution — Glutamine is an essential amino acid. It will be provided in a powder form. It will be dissolved in at least 8 ounces of hot or cold liquid. It can also be mixed with a soft food such as pudding, applesauce, or yogurt. Then it will be Stirred and then eaten or drunken The Glutamine will be as an add on to the Standard of care
  Other Names: L-Glutamine Powder
  Arms: cases
Other: Standard of care — Hydroxyurea 15-25 mg per kg per day and/ or blood transfusion therapy
  Arms: control

SUMMARY:
Prospective phase IV interventional open label randomized controlled trial to assess safety and efficacy of glutamine in preventing vaso-occlusive crisis (VOC) episodes in sickle cell pediatrics and adolescents' patients

DETAILED DESCRIPTION:
Vaso-occlusive crisis (VOC) episodes are considered to be the cause of 95% of hospitalizations for sickle cell disease (SCD) patients. Prior studies have described pain management in SCD patients with poor outcomes in the short term and decreased quality of life in patients over the long term.

Although that L-glutamine has been recently approved by the FDA for the prevention of acute complications in sickle cell disease. However, there are many gaps in our understanding of its therapeutic implications in SCD. This study will assess the safety and efficacy of glutamine in preventing vaso-occlusive crisis (VOC) episodes in sickle cell pediatrics and adolescents' patients

ELIGIBILITY:
Inclusion Criteria:

Children and adolescents diagnosed with sickle cell disease by haemoglobin electrophoresis and had at least two pain crises (no upper limit) documented during the previous year; a pain crisis is defined as pain leading to treatment with a parenteral administered narcotic or ketolac in an emergency department (ED) (or outpatient treatment centre) or during hospitalization.

Patients receiving hydroxyurea at a fixed dose for at least 3 months before screening.

Exclusion Criteria:

Patients with sickle cell trait and other hemoglobinopathy.

-

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2024-01-07 (Actual)

PRIMARY OUTCOMES:
Number of pain crises | 24 weeks
  The number of pain crises will be counted from day 1 till end of treatment at week 24

SECONDARY OUTCOMES:
Changes in transcranial doppler | 24 weeks
  Calculate the change in transcranial doppler (TCD) time-averaged mean of the maximum velocity (TAMMV) arterial cerebral blood flow through the measuring of TCD flow velocity at day1 and at Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Fatma SE Ebeid, MD, Principal Investigator — Ain Shams University, Faculty of Medicine
Locations (2):
- Egypt (2):
  - Faculty of Medicine Ain Shams University Research Institute- Clinical Research Center, Cairo, Non-US
  - Ain Shams University, Cairo

IPD SHARING:
Plan to Share IPD: No